CLINICAL TRIAL: NCT06646419
Title: Boosting Regional Integration for COPD Care Through Guided Implementation and Audit of Post Exacerbation Transition Bundle: A Multicentre , Prospective, Cluster Randomization, Inteventional Clinical Study
Brief Title: Boosting Regional Integration for COP D Care Through Guided Implementation and Audit of Post Exacerbation Transition Bundle
Acronym: BRIDGE-COPD
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980L00025
Record Dates: First submitted 2024-08-29; First posted 2024-10-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Intervention is implemented at a hospital level and will change overall daily practice. The intervention is composed of 3 active components: 1) education on guideline led disease knowledge and transition bundle led management pathway, 2) standardized transition bundle implementation, 3) clinical audit.Education begins at nearly 4 weeks before first subject in and keep learning every 4 weeks.
  Standardized transition bundle will be implemented once the first round education is completed. Clinical audit takes up after first subject enrolled and implemented every 12 weeks.
- Control group: The control group will maintain the current usual care practice.

SUMMARY:
This is a cluster randomized interventional study. Intervention is implemented at a hospital level and will change overall daily practice. 36 county level hospitals are r an domized to the intervention group or control group at the ratio of 2:1 . Total subjects is 1368 and a size of 38 per hospital .

DETAILED DESCRIPTION:
The intervention is composed of 3 active components: 1) education on guideline led disease knowledge and transition bundle led management pathway, 2) standardized transition bundle implementation, 3) clinical audit.

Education begins at nearly 4 weeks before first subject in and keep learning every 4 weeks.Standardized transition bundle will be implemented once the first round education is completed. Clinical audit takes up after first subject enrolled and implemented every 12 weeks.The control group will maintain the current usual care practice. Eligible patients will be recruited in both groups and will be followed up every 12 weeks for 48 weeks.

Eligible consented patients will be enrolled consecutively to minimize selection bias. In order to achieve the purpose of continuous enrollment, all patients who visit the outpatient clinic,emergency room, and hospitalized due to exacerbation of COPD will be screened, including newly diagnosed patients or those who have bee n treated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD (post- bronchodilator FEV1/FVC < 0.7)
* 40~80 years
* CAT≥10
* At least two moderate or at least one severe exacerbation history in past 1 year
* Able to sign informed consent

Exclusion Criteria:

* Continuous triple inhalation therapy for ≥6 months at baseline (include single inhaler and multiple inhalers)
* Stable COPD (symptom such as cough, sputum and shortness of breath are mild or stable, clinical condition has basically returned to pre-exacerbation)
* Comorbidities require/contraindicate long-term use of glucocorticoid treatment: asthma, interstitial lung disease, sarcoidosis, cystic fibrosis, active tuberculosis recurrent aspiration pneumonia ect.
* Serious comorbidities threaten to life expected survival time no more than 1 year: severe heart disease, severe chronic liver, severe kidney disease, cerebrovascular disease with long-term bed rest and malignant tumours ect.
* Not living in the healthcare area
* Patients currently participating in any other interventional studies

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population in this study are in the hospital exacerbation COPD patients with high risk of future exacerbation. Exacerbation COPD is defined as an event characterized by dyspnea and/or cough and sputum that worsen over <14 days. Exacerbation of COPD are often associated with increased local and systemic inflammation caused by airway infection, pollution, or other insults to the lungs.. Screening occurs when AECOPD identified in emergency room, respiratory outpatient clinic or inpatient department. Enrolment occurs when AECOPD treated for several days entering recovery period and transferring to home.
Sampling Method: Non-Probability Sample
Enrollment: 1368 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to CID. | week0-week48
  To evaluate the the impact of implementation and audit of transition bundle on clinically important deterioration (CID).

SECONDARY OUTCOMES:
Proportion of patients received long-acting maintenance inhalation with the percentage of days covered (PDC) ≥70%. | week 12, 24, 36 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment compliance.
Inhalation therapy consistency rate with guideline. | week 12, 24, 36 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment compliance.
Inhaler device compliance,measured by the score of Test of the adherence to inhalers( TAI ) questionnare. | week 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment compliance.
Correct operation rate of inhalation device. | week 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment compliance.
Patient satisfaction rate with treatment. | week 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment satisfaction.
Disease knowledge score of patients. | week 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on disease knowledge.
Proportion of patients received different categories of long-acting maintenance inhalation. | week 12, 24,36 and 48
  To evaluate the the impact of implementation and audit of transition bundle on treatment pattern.
Rate of moderate or severe exacerbation. | week 12, 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on exacerbation.
Rate of severe exacerbation. | week 12, 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on exacerbation.
Rate of cardiovascular events. | week 12, 24 and 48
  To evaluate the the impact of implementation and audit of transition bundle on cardiovascular events.
Change of CAT score. | week 0 to week 48
  To evaluate the the impact of implementation and audit of transition bundle on quality of life.
Percentage change of trough FEV1 and MMEF. | week 0 to week 48
  To evaluate the the impact of implementation and audit of transition bundle on PFT.

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - Research Site, Anyang
  - Research Site, Baise City
  - Research Site, Beijing
  - Research Site, Bijie
  - Research Site, Changsha
  - Research Site, Chenzhou
  - Research Site, Chifeng
  - Research Site, Chuzhou
  - Research Site, Deyang
  - Research Site, Fuyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jieyang
  - Research Site, Jining
  - Research Site, Jiujiang
  - Research Site, Kaiyuan
  - Research Site, Langfang
  - Research Site, Langzhong
  - Research Site, Leping
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Neijiang
  - Research Site, Qiannan
  - Research Site, Qujing
  - Research Site, Sanmenxia
  - Research Site, Shaoyang
  - Research Site, Suzhou
  - Research Site, Tengzhou
  - Research Site, Tieling
  - Research Site, Wenzhou
  - Research Site, Xiangtan
  - Research Site, Xiaogan
  - Research Site, Xinyang
  - Research Site, Yancheng
  - Research Site, Yichang
  - Research Site, Yuling
  - Research Site, Zaoyang

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. 'Yes' , indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/